CLINICAL TRIAL: NCT01107184
Title: A Clinical Study on the Effect of Remote Ischemic Conditioning on Atrial Fibrillation and Outcome After Coronary Artery Bypass Grafting
Brief Title: Remote Ischemic Conditioning and Atrial Fibrillation After Coronary Artery Bypass Grafting (CABG)
Acronym: RICO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, B Preckel, Prof. dr. B. Preckel, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NL 28041.018.09
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Atrial Fibrillation
Keywords: Remote ischemic conditioning; CABG surgery; Atrial fibrillation; Coronary Artery Bypass; Ischemic Preconditioning
MeSH Terms: conditions — Atrial Fibrillation | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Preconditioning (Experimental): The remote ischemic stimulus will be applied after induction of anaesthesia, but before cardiopulmonary bypass.
  Interventions: Procedure: Remote ischemic conditioning
- Postconditioning (Experimental): The remote ischemic stimulus during cardiopulmonary bypass.
  Interventions: Procedure: Remote ischemic conditioning
- Pre and postconditioning (Experimental): The remote ischemic stimulus will be applied twice, after induction of anaesthesia and during cardiopulmonary bypass.
  Interventions: Procedure: Remote ischemic conditioning
- Control (Sham Comparator)
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Patients will have a automated inflator cuff placed on the upper arm during surgery. The cuff will be used to induce fore arm ischemia by inflation to 200 mmHg for 3 x 5 minutes, interspersed with 5 minutes of no-inflation and thus reperfusion.
  Other Names: Remote ischemic preconditioning; Remote ischemic postconditioning
  Arms: Postconditioning; Pre and postconditioning; Preconditioning
Procedure: Sham — Patients will have a automated inflator cuff placed on the upper arm during surgery which will not be inflated.
  Arms: Control

SUMMARY:
Recent studies indicate that remote ischemic conditioning can protect the heart and other organs during cardiac surgery. The investigators aim to investigate whether such a stimulus can reduce the incidence of atrial fibrillation or other complications following coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective on-pump CABG surgery
* Informed consent

Exclusion Criteria:

* Prior cardiac surgery (Re-operations)
* Prior atrial fibrillation
* Use of class 1 or 3 anti arrhythmic medication or digoxin Use of intermittent aortic cross clamping during surgery
* Age <18 years
* Left ventricular ejection fraction ≤30%
* Serious pulmonary disease (resting pO2 <90% at room air)
* Renal failure (clearance <30 ml/min as calculated using the Modification of Diet in Renal Disease formula)
* Liver failure
* Use of the sulfonylurea derivative glibenclamide (this drug is known to block any preconditioning stimulus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2010-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Post-operative atrial fibrillation | 72 hours

SECONDARY OUTCOMES:
Major cardiovascular and cerebrovascular events | 3 months, 6 months, 1 year
  Major adverse events, i.e. death, acute coronary syndrome, stroke.
Length of stay | 1 week on avarage
  Duration of hospitalization and stay on the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Stef de Hert, Md, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, University of Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Derived] Brevoord D, Hollmann MW, De Hert SG, van Dongen EH, Heijnen BG, de Bruin A, Tolenaar N, Schlack WS, Weber NC, Dijkgraaf MG, de Groot JR, de Mol BA, Driessen AH, Momeni M, Wouters P, Bouchez S, Hofland J, Luthen C, Meijer-Treschan TA, Pannen BH, Preckel B. Effect of remote ischemic conditioning on atrial fibrillation and outcome after coronary artery bypass grafting (RICO-trial). BMC Anesthesiol. 2011 May 23;11:11. doi: 10.1186/1471-2253-11-11. PMID 21605453